CLINICAL TRIAL: NCT02571933
Title: Face Validity and Cross-Cultural Acceptability of the FPS-R in Cameroon
Acronym: FPS-RCam
Status: Completed | Type: Observational
Sponsor: Cameroon Baptist Convention Health (Other)
Collaborators: Carolinas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: IRB2015-04
Record Dates: First submitted 2015-09-29; First posted 2015-10-08 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Pain
Keywords: Pediatrics; Pain Scale; Faces Pain Scale - Revised; Cameroon
MeSH Terms: conditions — Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Grammar English: Patients who primarily speak Grammar English. Patients will answer the FPS-R in Grammar English both before and after administration of routine analgesia for pain (analgesia to be administered regardless of enrollment in study). Study participants will answer a series of questions - the cognitive interview - after second FPS-R to assess for ease of use and how well it is understood.
  Interventions: Other: Pre-treatment Faces Pain Scale - Revised; Other: Post-treatment Faces Pain Scale - Revised; Other: Cognitive interview
- Pidgin English: Patients who primarily speak Pidgin English. Patients will answer the FPS-R in Pidgin English both before and after administration of routine analgesia for pain (analgesia to be administered regardless of enrollment in study). Study participants will answer a series of questions - the cognitive interview - after second FPS-R to assess for ease of use and how well it is understood.
  Interventions: Other: Pre-treatment Faces Pain Scale - Revised; Other: Post-treatment Faces Pain Scale - Revised; Other: Cognitive interview
- French: Patients who primarily speak French. Patients will answer the FPS-R in French both before and after administration of routine analgesia for pain (analgesia to be administered regardless of enrollment in study). Study participants will answer a series of questions - the cognitive interview - after second FPS-R to assess for ease of use and how well it is understood.
  Interventions: Other: Pre-treatment Faces Pain Scale - Revised; Other: Post-treatment Faces Pain Scale - Revised; Other: Cognitive interview

INTERVENTIONS:
Other: Pre-treatment Faces Pain Scale - Revised — Patients will be asked to answer the Faces Pain Scale - Revised as an assessment of pain prior to standard analgesia dosing.
Other: Post-treatment Faces Pain Scale - Revised — Patients will be asked to answer the Faces Pain Scale - Revised 1-2 hours after receiving standard analgesia as an assessment of pain.
Other: Cognitive interview — Patients will answer a series of questions pertaining to the pain scale's ease of use, intuitive nature, and cultural appropriateness.

SUMMARY:
This study evaluates the face validity and cultural acceptability of the Faces Pain Scale - Revised in pediatric patients treated at Mbingo Baptist Hospital, Northwest Province, Cameroon. Participants from the four major language/cultural groups evaluated at the hospital with a complaint of pain will trial the Faces Pain Scale - Revised and then undergo cognitive interviewing to assess comprehension and clinical accuracy.

DETAILED DESCRIPTION:
Twelve to fifteen pediatric patients complaining of pain from each of the four primary language groups treated at Mbingo Baptist Hospital (Grammar English, Pidgin English, French, and Fulfulde) will be enrolled in the study. Each patient enrolled will trial the Faces Pain Scale - Revised (FPS-R) in his or her native tongue, before receiving standard analgesic treatment as ordered by the provider caring for the patient. One to two hours post analgesia, the patient will be reassessed and the FPS-R will be repeated. After completion of the second FPS-R, an audio-recorded cognitive interview will be performed by trained study personnel. These recordings will be transcribed into English and analyzed on a question-by-question basis to evaluate for themes pertaining to comprehension and understanding, ease of use, and reliability, within the different language groups. Enrollment in the study does not alter the routine pain management offered or received by patients. Rather, the FPS-R will be utilized on patients who are complaining of pain and who will be allocated to receive analgesia regardless of study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Children's Ward
* Complaint of pain

Exclusion Criteria:

* Coma
* Traumatic brain injury
* Glasgow Coma Scale (GCS) < 13
* Cognitive delay
* Narcotic/opioid dependency

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Study population encompasses the four primary language-defined cultural groups that present to Mbingo Baptist Hospital. Goal of 12-15 pediatric patients per cohort (Grammar English, Pidgin English, French, and Fulfulde speaking), who have pain as part of their presenting complaint.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Face validity of pain scale as assessed by cognitive interview probes | Through study completion, an average of 3 months
  Detailed qualitative review of cognitive interview probes with question-by-question analysis of transcribed cognitive interviews to assess for basic comprehension and appropriate use of the FPS-R.
Face validity of pain scale as assessed by FPS-R results | Through study completion, an average of 3 months
  Detailed review of the FPS-R answers provided by patients in the context of their illness/injury.
Cultural acceptability of pain scale as assessed by cognitive interview probes | Through study completion, an average of 3 months
  Question-by-question analysis and review of transcribed cognitive interviews to search for thematic responses that correspond to cultural understanding and ease of use.

CONTACTS AND LOCATIONS:
Overall Officials: James R Young, MD, Principal Investigator — Carolinas Medical Center
Locations (1):
- Mbingo Baptist Hospital, Mbingo, Northwest Province, Cameroon

REFERENCES:
- [Background] Beatty PC, Willis BG, "Research synthesis: the practice of cognitive interviewing. Public Opin Q, 2007, 71:287-311
- [Background] Cartledge P, et al, "A pilot acceptability study of the Paediatric Faces Pain Scale among adults attending a sub-Saharan hospice. PCAU J Palliat Care 2005, 7:14-18
- [Background] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329
- [Background] Huang KT, Owino C, Vreeman RC, Hagembe M, Njuguna F, Strother RM, Gramelspacher GP. Assessment of the face validity of two pain scales in Kenya: a validation study using cognitive interviewing. BMC Palliat Care. 2012 Jul 10;11:5. doi: 10.1186/1472-684X-11-5. PMID 22512923
- [Background] Jensen MP, Karoly P, Braver S. The measurement of clinical pain intensity: a comparison of six methods. Pain. 1986 Oct;27(1):117-126. doi: 10.1016/0304-3959(86)90228-9. PMID 3785962
- [Background] Miro J, Huguet A. Evaluation of reliability, validity, and preference for a pediatric pain intensity scale: the Catalan version of the faces pain scale--revised. Pain. 2004 Sep;111(1-2):59-64. doi: 10.1016/j.pain.2004.05.023. PMID 15327809
- [Background] Newman CJ, Lolekha R, Limkittikul K, Luangxay K, Chotpitayasunondh T, Chanthavanich P. A comparison of pain scales in Thai children. Arch Dis Child. 2005 Mar;90(3):269-70. doi: 10.1136/adc.2003.044404. PMID 15723913
- [Background] Stinson JN, Kavanagh T, Yamada J, Gill N, Stevens B. Systematic review of the psychometric properties, interpretability and feasibility of self-report pain intensity measures for use in clinical trials in children and adolescents. Pain. 2006 Nov;125(1-2):143-57. doi: 10.1016/j.pain.2006.05.006. Epub 2006 Jun 13. PMID 16777328
- [Background] Tomlinson D, von Baeyer CL, Stinson JN, Sung L. A systematic review of faces scales for the self-report of pain intensity in children. Pediatrics. 2010 Nov;126(5):e1168-98. doi: 10.1542/peds.2010-1609. Epub 2010 Oct 4. PMID 20921070
- [Background] Willis GB, Cognitive Interviewing: a tool for improving questionnaire design. Thousand Oaks, Sage Publications, 2005.
- [Background] Woolley ME, Bowen GL, Bowen NK. Cognitive Pretesting and the Developmental Validity of Child Self-Report Instruments: Theory and Applications. Res Soc Work Pract. 2004 May;14(3):191-200. doi: 10.1177/1049731503257882. PMID 21709820